CLINICAL TRIAL: NCT04319536
Title: Integrated Genetic and Functional Analysis of the Female Microbiome in a Flemish Cohort
Acronym: Isala
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Professor, Universiteit Antwerpen
Other Study IDs: B300201942076
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Vaginal Microbiome; Skin Microbiome; Saliva Microbiome
Keywords: Metagenomic sequencing; vaginal microbiome; skin microbiome; saliva microbiome; large-scale self-sampling cohort; Microbiota; Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbial DNA will be analysed from swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — self-sampling

SUMMARY:
The aim of the project is to improve our knowledge on the stability and temporal dynamics of the Flemish female microbiome (vagina, skin and saliva) in relation to different lifestyle factors and environmental conditions and to establish certain individual and social risk factors that can influence the healthy microbiome. Therefore, microbial DNA from swabs will be isolated via commercially available DNA extraction kits, followed by Illumina MiSeq sequencing in order to identify the microbial species present in these samples. Special attention will go to microbial species that are overrepresented in the healthy populations as potential health promoting microbes (i.e. probiotics).

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations involves healthy women from 18 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Differences in microbial communities colonizing the vagina, skin and saliva between healthy individuals measured with Illumina MiSeq | up to 5 years
  After metagenomic shotgun and amplicon sequencing with the Illumina MiSeq, bio-informatic tools will be used to analyse taxonomic and functional data. The investigators will specifically screen for health-promoting and pathogenic taxa that can be associated with specific environmental conditions and lifestyle factors. Additionally, the investigators will pay attention to the dominant members of the vaginal bacterial community (i.e. beneficial microbes such as lactic acid bacteria).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp and University Hospital Antwerp, Antwerp, Belgium